CLINICAL TRIAL: NCT07151742
Title: Investigation of the Effects of Intradialytic Combined Exercises on Dialysis Parameters and Muscle Oxygenation in Sarcopenic Hemodialysis Patients
Brief Title: Effects of Intradialytic Exercise on Muscle Oxygenation and Dialysis Adequacy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Beyza DAL KOYUNCUOĞLU, Research Assistant, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-123
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease, Stage 5; Sarcopenia
Keywords: Hemodialysis; sarcopenia; Intradialytic exercise; muscle oxygenation; Dialysis Parameters
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with two parallel groups. A total of 40 eligible patients undergoing maintenance hemodialysis will be enrolled and randomly assigned in a 1:1 ratio to either the intervention group (n=20), receiving a 12-week intradialytic combined exercise program, or the control group (n=20), receiving routine hemodialysis care. Randomization will be performed using a computer-generated sequence, and allocation will be parallel without masking, as the intervention cannot be blinded.
Who Masked: Participant
Masking Description: Participants were aware of their group assignment (exercise or routine care) due to the nature of the intervention. Neither researchers nor outcome assessors were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants in this arm will receive a 12-week intradialytic combined exercise program, performed three times per week during the first two hours of hemodialysis. Each session will begin with a 10-minute warm-up and end with a 10-minute cool-down (stretching and breathing exercises).
  Aerobic component: Supine cycling using a portable ergometer at 45-70% of maximum heart rate, monitored with pulse oximetry and Borg scale, progressively increased every 1-2 weeks.
  Resistance component: Exercises with elastic bands and ankle weights targeting major upper and lower extremity muscle groups (non-fistula arm). Performed in 2 sets of 8-12 repetitions, with progressive loading based on ACSM guidelines.
  All sessions will be supervised by trained physiotherapists and dialysis staff to ensure safety and adherence
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Control Group (No Intervention): Participants in this arm will continue routine hemodialysis care for 12 weeks. In addition, they will receive general recommendations for breathing and posture exercises to be performed outside dialysis sessions. These exercises will not be structured or supervised, and no additional training program will be provided during dialysis

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Participants in this arm will receive a 12-week intradialytic combined exercise program, performed three times per week during the first two hours of hemodialysis. Each session will begin with a 10-minute warm-up and end with a 10-minute cool-down (stretching and breathing exercises).
  Aerobic component: Supine cycling using a portable ergometer at 45-70% of maximum heart rate, monitored with pulse oximetry and Borg scale, progressively increased every 1-2 weeks.
  Resistance component: Exercises with elastic bands and ankle weights targeting major upper and lower extremity muscle groups (non-fistula arm). Performed in 2 sets of 8-12 repetitions, with progressive loading based on ACSM guidelines.
  All sessions will be supervised by trained physiotherapists and dialysis staff to ensure safety and adherence
  Other Names: intradialytic exercise
  Arms: Exercise Group

SUMMARY:
This randomized controlled trial will evaluate the effects of a 12-week intradialytic combined exercise program, consisting of aerobic and resistance training, in patients with stage 5 chronic kidney disease receiving maintenance hemodialysis. Sarcopenia, a progressive loss of muscle mass and strength, is common in this population due to chronic disease burden and the sedentary nature of dialysis sessions. The intervention group will perform structured exercise three times per week during the first two hours of dialysis, while the control group will continue routine dialysis care without exercise.

The primary aim is to investigate whether intradialytic exercise can improve dialysis adequacy and muscle oxygenation, and reduce sarcopenia severity. Secondary objectives include evaluating changes in physical performance, muscle strength, fatigue levels, and health-related quality of life. Approximately 40 participants will be randomized into intervention and control groups. Outcomes will be assessed through clinical measurements, functional tests, and patient-reported questionnaires before and after the intervention period.

DETAILED DESCRIPTION:
Sarcopenia is a progressive loss of skeletal muscle mass and strength, associated with physical disability, poor quality of life, and increased mortality risk. Although commonly linked to aging, sarcopenia may also develop as a secondary condition in patients with chronic kidney disease (CKD) due to malnutrition, low physical activity, or treatment-related catabolism. In individuals undergoing hemodialysis, protein catabolism, inflammation, and nutrient loss are accelerated, further contributing to sarcopenia. Prolonged dialysis sessions also enforce sedentary behavior, exacerbating physical decline.

Exercise interventions have been shown to delay sarcopenia progression, improve functional capacity, and support survival. Intradialytic exercise, performed during dialysis sessions, offers practical advantages as it is time-efficient, conducted under medical supervision, and associated with better adherence compared to exercise outside dialysis. Combined programs involving both aerobic and resistance training are particularly effective in improving dialysis adequacy, reducing fatigue, and supporting muscle maintenance.

Muscle oxygenation plays an important role in sarcopenia. Factors such as oxidative stress, mitochondrial dysfunction, and impaired circulation can reduce oxygen delivery and utilization, leading to muscle weakness and atrophy. Hemodialysis itself alters microcirculation and oxygenation, negatively affecting muscle recovery. Near-infrared spectroscopy (NIRS) enables non-invasive monitoring of muscle oxygenation and has demonstrated that exercise interventions can improve tissue oxygenation parameters.

This randomized controlled trial will investigate the effects of a 12-week intradialytic combined exercise program-including aerobic and resistance training-on dialysis adequacy, muscle oxygenation, and sarcopenia severity in patients with CKD undergoing maintenance hemodialysis. Secondary outcomes will include physical performance, fatigue, and health-related quality of life.

The study will be conducted at Kadıköy Dialife Ata Dialysis Center in Istanbul, Turkey. A total of 40 participants aged 18-65 with stage 5 CKD on maintenance hemodialysis for at least one year, and diagnosed with sarcopenia according to EWGSOP2 criteria, will be enrolled. Participants will be randomly assigned to either an exercise group or a control group.

Intervention group: Participants will receive a 12-week intradialytic combined exercise program performed three times per week during the first two hours of dialysis sessions. Aerobic training will consist of supine cycling with a portable ergometer at 45-70% of maximum heart rate, adjusted progressively and monitored with pulse oximetry and the Borg scale. Resistance training will include exercises with elastic bands and ankle weights targeting upper and lower extremities, performed as 2 sets of 8-12 repetitions with progressive load increments according to ACSM guidelines. Each session will also include a 10-minute warm-up and cool-down with stretching and breathing exercises.

Control group: Participants will receive routine hemodialysis care without structured exercise. After completion of the study, the exercise program will be offered to this group.

Safety monitoring: Exercise intensity will be individualized. Sessions will be interrupted in cases of chest pain, dizziness, hypotension, severe fatigue, or excessive perceived exertion. Continuous monitoring of heart rate, blood pressure, and oxygen saturation will be conducted.

Primary outcomes will include dialysis adequacy (Kt/V, URR) and muscle oxygenation (SmO₂) assessed by NIRS. Secondary outcomes will include handgrip strength, body composition, peripheral muscle strength, the 6-minute walk test (6MWT), the Short Physical Performance Battery (SPPB), fatigue severity, quality of life (KDQOL-36), and selected laboratory parameters.

Statistical analysis will be performed using appropriate parametric or non-parametric tests according to data distribution. Significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Diagnosed with stage 5 chronic kidney disease (end-stage renal disease) according to GFR, undergoing maintenance hemodialysis for at least 1 year

Diagnosed with sarcopenia based on EWGSOP2 (2018) criteria

Able to read and write

Cooperative and able to follow instructions

Voluntary participation with written informed consent

Exclusion Criteria:

Presence of orthopedic or neurological disorders affecting mobility or exercise capacity

Uncontrolled diabetes mellitus or uncontrolled hypertension

Untreated intradialytic hypotension

Heart failure

Unstable angina

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Oxygen Saturation (SmO₂, %) | Baseline and after 12 weeks
  Muscle oxygen saturation (SmO₂) will be measured non-invasively using near-infrared spectroscopy (Moxy device) placed over the vastus lateralis muscle. Average SmO₂ values will be recorded at rest, during a 6-minute walk test, and during post-exercise recovery to assess local oxygen delivery and utilization.
Total Hemoglobin Concentration | Baseline and after 12 weeks
  Total hemoglobin concentration will be measured non-invasively using near-infrared spectroscopy (Moxy device) placed over the vastus lateralis muscle. Values will be recorded at rest, during a 6-minute walk test, and during post-exercise recovery to evaluate local oxygen delivery and utilization.
Dialysis Adequacy - Kt/V | Baseline and after 12 weeks
  Dialysis adequacy will be assessed using pre- and post-dialysis blood urea nitrogen (BUN) levels. Kt/V will be calculated to evaluate the effectiveness of hemodialysis treatment. Higher values indicate better dialysis efficiency.
Dialysis Adequacy - Urea Reduction Ratio | Baseline and after 12 weeks
  Dialysis adequacy will be assessed using pre- and post-dialysis blood urea nitrogen (BUN) levels. Urea Reduction Ratio (URR) will be calculated to evaluate the effectiveness of hemodialysis treatment. Higher values indicate better dialysis efficiency.

SECONDARY OUTCOMES:
Handgrip Strength | Baseline
  Grip strength will be measured using a Jamar dynamometer according to American Society of Hand Therapists' standard procedures. Three attempts will be recorded for both dominant and non-dominant hands, and the maximum value (kg) will be used.
Fat-Free Mass Index | Baseline
  Fat-free mass index (FFMI, kg/m²) will be assessed by Bioelectrical Impedance Analysis (BIA).
Peripheral Muscle Strength | Baseline and after 12 weeks
  Muscle strength of major upper and lower limb groups will be assessed using a digital dynamometer. Upper limb measurements (shoulder and elbow flexors) will be performed on the non-fistula arm, while lower limb measurements (hip flexors and knee extensors) will be performed bilaterally.
Six-Minute Walk Test (6MWT) | Baseline and after 12 weeks
  Muscle oxygenation measurements will be taken at rest, during a 6-minute walk test (6MWT), and during recovery. The 6MWT will serve solely as a standardized protocol for eliciting muscle activity during NIRS monitoring, not as an independent functional outcome.
Short Physical Performance Battery (SPPB) | Baseline and after 12 weeks
  Physical performance will be assessed by SPPB, including sit-to-stand test, balance tests, and gait speed. Scores range from 0-12, with lower scores indicating poorer performance.
Fatigue Severity Scale (FSS) | Baseline and after 12 weeks
  Patient-reported fatigue will be assessed using the FSS, a 9-item Likert-type questionnaire. Higher mean scores indicate greater fatigue severity.
Kidney Disease Quality of Life (KDQOL-36) | Baseline and after 12 weeks
  Health-related quality of life will be measured with the KDQOL-36, covering symptom burden, effects and burden of kidney disease, and physical/mental health components. Higher scores reflect better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadıköy Ata Dialysis Center, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because data sharing was not included in the informed consent process.

REFERENCES:
- [Background] Yu MD, Zhang HZ, Zhang Y, Yang SP, Lin M, Zhang YM, Wu JB, Hong FY, Chen WX. Relationship between chronic kidney disease and sarcopenia. Sci Rep. 2021 Oct 15;11(1):20523. doi: 10.1038/s41598-021-99592-3. PMID 34654871
- [Background] Umakanthan M, Li JW, Sud K, Duque G, Guilfoyle D, Cho K, Brown C, Boersma D, Gangadharan Komala M. Prevalence and Factors Associated with Sarcopenia in Patients on Maintenance Dialysis in Australia-A Single Centre, Cross-Sectional Study. Nutrients. 2021 Sep 20;13(9):3284. doi: 10.3390/nu13093284. PMID 34579163
- [Background] Shen S, Liao Q, Lyu P, Wang J, Lin L. Myricanol prevents aging-related sarcopenia by rescuing mitochondrial dysfunction via targeting peroxiredoxin 5. MedComm (2020). 2024 Jun 12;5(6):e566. doi: 10.1002/mco2.566. eCollection 2024 Jun. PMID 38868327
- [Background] Shahar S, Kamaruddin NS, Badrasawi M, Sakian NI, Abd Manaf Z, Yassin Z, Joseph L. Effectiveness of exercise and protein supplementation intervention on body composition, functional fitness, and oxidative stress among elderly Malays with sarcopenia. Clin Interv Aging. 2013;8:1365-75. doi: 10.2147/CIA.S46826. Epub 2013 Oct 9. PMID 24143082
- [Background] Savaş, S. (2015). Sarkopeniden korunma. Ege Tıp Dergisi, 54(0), 29-36. https://doi.org/10.19161/etd.344148
- [Background] Sanchez-Tocino ML, Gonzalez-Parra E, Miranda Serrano B, Gracia-Iguacel C, de-Alba-Penaranda AM, Lopez-Gonzalez A, Garcia Olegario M, Ortiz A, Mas-Fontao S. Evaluation of the impact of an intradialytic exercise programme on sarcopaenia in very elderly haemodialysis patients. Clin Kidney J. 2022 Feb 15;15(8):1514-1523. doi: 10.1093/ckj/sfac046. eCollection 2022 Aug. PMID 35892024
- [Background] Sabatino A, Cuppari L, Stenvinkel P, Lindholm B, Avesani CM. Sarcopenia in chronic kidney disease: what have we learned so far? J Nephrol. 2021 Aug;34(4):1347-1372. doi: 10.1007/s40620-020-00840-y. Epub 2020 Sep 2. PMID 32876940
- [Background] Pipili C, Grapsa E, Tripodaki ES, Ioannidou S, Manetos C, Parisi M, Nanas S. Changes in skeletal muscle microcirculation after a hemodialysis session correlates with adequacy of dialysis. Int J Nephrol Renovasc Dis. 2015 Jun 8;8:59-64. doi: 10.2147/IJNRD.S68639. eCollection 2015. PMID 26089698
- [Background] Pender D, McGowan E, McVeigh JG, McCullagh R. The Effects of Intradialytic Exercise on Key Indices of Sarcopenia in Patients With End-stage Renal Disease: A Systematic Review of Randomized Controlled Trials. Arch Rehabil Res Clin Transl. 2023 Jan 13;5(1):100252. doi: 10.1016/j.arrct.2022.100252. eCollection 2023 Mar. PMID 36968168
- [Background] Moriyama Y, Hara M, Aratani S, Ishikawa H, Kono K, Tamaki M. The association between six month intra-dialytic resistance training and muscle strength or physical performance in patients with maintenance hemodialysis: a multicenter retrospective observational study. BMC Nephrol. 2019 May 16;20(1):172. doi: 10.1186/s12882-019-1375-1. PMID 31096932
- [Background] McManus CJ, Collison J, Cooper CE. Performance comparison of the MOXY and PortaMon near-infrared spectroscopy muscle oximeters at rest and during exercise. J Biomed Opt. 2018 Jan;23(1):1-14. doi: 10.1117/1.JBO.23.1.015007. PMID 29368457
- [Background] Krase AA, Terzis G, Giannaki CD, Stasinaki AN, Wilkinson TJ, Smith AC, Zorz C, Karatzaferi C, Stefanidis I, Sakkas GK. Seven months of aerobic intradialytic exercise training can prevent muscle loss in haemodialysis patients: an ultrasonography study. Int Urol Nephrol. 2022 Feb;54(2):447-456. doi: 10.1007/s11255-021-02931-6. Epub 2021 Jun 28. PMID 34184202
- [Background] Hu H, Wu C, Kwok JYY, Ho MH, Chau PH, Lok KYW, Choi EPH. Effects of Different Exercises on Physical Function, Dialysis Adequacy, and Health-Related Quality of Life in Maintenance Hemodialysis Patients: A Systematic Review and Network Meta-Analysis. Am J Nephrol. 2023;54(9-10):379-390. doi: 10.1159/000532109. Epub 2023 Aug 3. PMID 37536298
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Almushayt SJ, Hussain S, Wilkinson DJ, Selby NM. A Systematic Review of the Acute Effects of Hemodialysis on Skeletal Muscle Perfusion, Metabolism, and Function. Kidney Int Rep. 2019 Dec 30;5(3):307-317. doi: 10.1016/j.ekir.2019.12.012. eCollection 2020 Mar. PMID 32154452
- See also: Related Info — https://link.springer.com/article/10.1007/s11255-021-02931-6